CLINICAL TRIAL: NCT01299298
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation, Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Single Doses of Mipomersen Administered Subcutaneously to Japanese Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Single Doses of Mipomersen in Japanese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MIPO3700710; 2010-021948-18 (EudraCT Number)
Record Dates: First submitted 2011-02-09; First posted 2011-02-18 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — mipomersen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mipomersen (Experimental): 50 mg (cohort A), 100mg (cohort B) or 200mg (cohort C) SC single dose
  Interventions: Drug: mipomersen
- placebo (Placebo Comparator): 50 mg (cohort A), 100mg (cohort B) or 200mg (cohort C) SC single dose
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: mipomersen — 50 mg (cohort A), 100mg (cohort B) or 200mg (cohort C) subcutaneous (SC) single dose of study drug
  Other Names: ISIS 301012
  Arms: mipomersen
Drug: placebo — 50 mg (cohort A), 100mg (cohort B), or 200mg (cohort C) subcutaneous (SC) single dose of study drug
  Arms: placebo

SUMMARY:
This Phase 1 study is being conducted to evaluate 3 increasing subcutaneous (SC) doses (50, mg, 100 mg or 200mg) of mipomersen in Japanese healthy volunteers. Eligible subjects will receive a single study injection of either mipomersen or placebo. Subjects will be enrolled into 1 of 3 treatment cohorts (Cohorts A, B, and C) in a dose-escalation design. Dose-escalation will proceed only if there is an acceptable safety profile from the previous dosing level.

ELIGIBILITY:
Inclusion Criteria:

* First generation Japanese (born in Japan of Japanese parents and Japanese grandparents), lived no more than 5 years outside of Japan, with no significant change in lifestyle or habits, including diet, while living outside of Japan.
* Surgically sterile, abstinent or subject or partner compliant with acceptable contraceptive during and 24 weeks after the last study drug dose
* Body weight >50 kg and body mass index between 18 and 30 kg/m2 inclusive

Exclusion Criteria:

* Clinically significant cardiovascular, pulmonary, hepatic, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, infectious, or psychiatric disease
* Clinically significant abnormal findings on the physical examination, ECG, blood pressure, heart rate, medical history, or clinical laboratory results at Screening or before dosing
* Positive test for human immunodeficiency virus (HIV), hepatitis B or C.
* High sensitivity C-reactive protein (hsCRP) >5 mg/L
* History of or current malignancy (with the exception of basal or squamous cell carcinoma of the skin if adequately treated and no recurrence for > 1 year)
* Evidence of acute or ongoing chronic inflammatory condition or infection
* History of rash, impetigo, or drug allergies
* Alcohol and/or drug abuse
* Smoking more than 10 cigarettes per day
* Planned dental work up to and including Day 8 procedures
* Treatment with another investigational drug, biological agent, or device within 4 weeks of Screening or 5 half-lives of the study agent, whichever is longer
* Use of prescribed medications within 4 weeks or over-the counter medications (including dietary supplements and herbal remedies) within 14 days before the first study drug dose, or use of any concomitant medications (prescribed or over the counter) through Day 8 of the study without Investigator and Sponsor approval. Vaccinations are not allowed beginning 3 weeks prior to the first dose of study drug until completion of the safety follow-up period
* Previous exposure to oligonucleotide-based drug therapy
* Donated 50 to 499 mL of blood within 30 days prior to consent, or >499 mL within 60 days

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Baseline up to Day 36 Post-Treatment
  plasma PK parameters
Time to maximal concentration (Tmax) | Baseline up to Day 36 Post-Treatment
  plasma PK parameters
Area Under the Curve (AUC) | Baseline up to Day 36 Post-Treatment
  plasma PK parameters

SECONDARY OUTCOMES:
Number of Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 36 Post-Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- FOCUS Clinical Drug Development GmbH, Stresemannallee 6, Neuss, Germany